CLINICAL TRIAL: NCT01565252
Title: Assessment of the Effect of n-3(Omega 3) Fortified Egg Compared to Omega-6 Israeli Regular Egg on Metabolic, Inflammation and Other Physiologic Parameters Prospective, Crossover, Compared Study in Healthy Subjects
Brief Title: Assessment of the Effect of n-3(Omega 3) Fortified Egg in Healthy Subjects
Acronym: PisNShMiGSL-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre singer, Professor, MD, Rabin Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6445
Record Dates: First submitted 2012-03-09; First posted 2012-03-28 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Volunteers
Keywords: Egg,Omega 3, Omega 6

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage 1 (No Intervention): Dietary regimens:
  Stage1 - all participants (N=20) in first stage will receive two regular (high n-6 PUFA) hard-boiled eggs/day at breakfast for a three weeks period for each participant.
- Stage 2 (Experimental): Stage 2 will be conduct after 3 weeks for wash-out with no eggs. All participants(N=20) in second stage will receive two high n-3 PUFA hard-boiled eggs/day at breakfast for a three weeks period for each participant.
  Interventions: Dietary Supplement: eggs enriched Omega-3

INTERVENTIONS:
Dietary Supplement: eggs enriched Omega-3 — In second stage participants will receive two Omega-3 enriched hard-boiled eggs/day at breakfast for a three weeks period for each participant.
  Arms: Stage 2

SUMMARY:
Study Rationale:

As epidemiological research has shown negative effects of high egg consumption on increased all-cause mortality and diabetes and on diabetes outcomes, and egg modification may modulate their effects on diseases risks, it is important to test the effect of eggs with different composition on markers associated with dyslipidemia, dysglycemia and inflammation.

The aim of this study is to assess the effect of n-3PUFA (Omega 3) fortified egg compared to omega-6 Israeli regular egg on metabolic, inflammation and other physiologic parameters.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

First endpoint:

To assess the effect of high n-3 PUFA (Omega 3) egg, as compared to regular- high n-6 PUFA (Omega 6) Israeli egg, on glycemic levels after night fasting and post prandial of 2 egg breakfast test meal.

Secondary endpoint:

To compare the effect of high n-3 PUFA fortified egg versus high n-6 PUFA (Regular) egg on measures associated with CVD risks including: CRP, LDL oxidation, MDA, post prandial Flow mediated dilatation (FMD), liver enzymes, and blood lipids and lipoproteins, and further blood chemistry measures.

Third endpoint:

To assess the influence of n-3 Egg on erythrocytes fatty acid profile.

Study design: Prospective, Crossover, Compared Study Study population: 20 Healthy subjects

Study Methods:

Subjects will complete two study stages. In first stage study participants will get 3 weeks regimen including 2 Regular, Israeli (high n-6 Pufa) eggs/day.

In second stage after 3 weeks washout without eggs, study participants will get 3 weeks regimen with 2 high n-3Pufa eggs/day.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men volunteers (age 18-45 years)
2. BMI 23-28

Exclusion Criteria:

1. Use of lipid-modifying medications or nutritional supplements
2. Known malignancy
3. Allergy to eggs or other materials use in the experiment
4. Substance abuse (including alcohol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Glycemic levels | before meal and 30 and 60 minutes after meal
  Pre- and Post-prandial (before meal and 30 and 60 minutes after meal) blood glucose test

SECONDARY OUTCOMES:
Fatty Acid Composition | Study Days:1,21,43 and 63
  ω3 incorporation into blood cell membranes(RBC)
C-Reactive protein | Study Days:1, 21, 43 and 63
  measures associated with CVD (Cardiovascular disease) risks
MDA(Malondialdehyde) | Study days: 1,21,43 and 63
  Measures associated with CVD (Cardiovascular disease) risks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Professor,MD, Principal Investigator — ICU dep't, Institute for Nutrition Research, Rabin MC; Niva Shapiro, Ph.D.,R.D., Study Chair — Institute for Nutrition Research, Rabin MC; Milana Grinev, Study Coordinator, Study Director — ICU dep't, Institute for Nutrition Research, Rabin MC
Locations (1):
- Rabin Medical Center, Campus Beilinson, Petah Tikva, Petach Tikva, Israel